CLINICAL TRIAL: NCT06302322
Title: Influence of Mucosal Tissue Height on Implant Crestal Bone Stability: A Longitudinal 10-year Cohort Study
Brief Title: Long-term Follow up of Mucosal Tissue Height Influence on Peri-implant Bone Levels.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, German O. Gallucci, Associate Professor and Chair Department of Restorative Dentistry and Biomaterials Sciences, Harvard Medical School (HMS and HSDM)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 158200-07-512-149
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Edentulous Alveolar Ridge
Keywords: dental implant; phenotype; mucosal tissues; mucosal tissue augmentation; vertical soft tissue height; bone resorption; bone remodeling; bone formation
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Natural Thin Gums (Experimental)
  Interventions: Procedure: Thin Tissues
- Natural Thick Gums (Experimental)
  Interventions: Procedure: Thick Tissues
- Surgically augmented Thin Gums (Experimental)
  Interventions: Procedure: Surgically augmented thin tissues

INTERVENTIONS:
Procedure: Thin Tissues — Patients with thin tissues received implants 10 years ago and are now followed up after 10 years.
  Arms: Natural Thin Gums
Procedure: Thick Tissues — Patients with thick tissues received implants 10 years ago and are now followed up after 10 years.
  Arms: Natural Thick Gums
Procedure: Surgically augmented thin tissues — Patients with thin tissues received soft tissue augmentation and implants 10 years ago and are now followed up after 10 years.
  Arms: Surgically augmented Thin Gums

SUMMARY:
Our study looks into how the thickness of the gum tissue affects the health of the bone around dental implants over ten years. We include 59 people and divide them into three groups based on their gum tissue thickness. Some have naturally thin gums, some have thin gums that were made thicker with a special procedure, and some already had thick gums. We try to find out if having thicker gums, whether naturally or through enhancement, can help keep the bone around dental implants healthy in the long run.

DETAILED DESCRIPTION:
The protocol of our study focuses on understanding the impact of gum tissue thickness on the stability of the bone surrounding dental implants over a period of ten years. We enroll 59 participants and categorize them based on their initial gum thickness. The study groups included participants with naturally thin gums, participants whose thin gums were surgically enhanced with an allogenic tissue matrix to increase thickness, and participants with naturally thick gums. We monitore the bone levels around the implants using X-rays at baseline and annually, assessing any changes in bone health and stability. Our objective is to determine if and how the thickness of gum tissue influences long-term bone preservation around dental implants, aiming to provide insights into better implant care and outcomes.

ELIGIBILITY:
The inclusion criteria for the study were individuals aged 18 years or older, generally healthy with no medical contraindications for implant surgery, missing teeth in the lower jaw posterior area, at least 6 mm bone width, healthy soft tissue, at least 2 mm keratinized gingiva buccally and lingually, no bone augmentation procedures before or during implant placement, and a signed informed consent form. The exclusion criteria included poor oral hygiene, history of uncontrolled periodontitis, smoking, diabetes, alcoholism, and medication influencing healing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Crestal Bone Levels | 10 year follow up
  Assessment of changes in crestal bone level (CBL)

SECONDARY OUTCOMES:
PPD | 10 year follow up
  Pocket probing depth
BOP | 10 year follow up
  Bleeding on Probing
PI | 10 year follow up
  Plaque Index

CONTACTS AND LOCATIONS:
Locations (1):
- VIC Clinic, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
We plan to make de-identified individual participant data (IPD) from our study on dental implant techniques available to other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Puisys A, Linkevicius T. The influence of mucosal tissue thickening on crestal bone stability around bone-level implants. A prospective controlled clinical trial. Clin Oral Implants Res. 2015 Feb;26(2):123-9. doi: 10.1111/clr.12301. Epub 2013 Dec 9. PMID 24313250